CLINICAL TRIAL: NCT00243113
Title: Multi-Institutional Phase II Study of Weekly Docetaxel and Concurrent Radiotherapy for Laryngeal and Hypopharyngeal Cancer in the Group of Elderly and/or Patients With Medical Illness
Brief Title: Docetaxel and Radiation Therapy in Treating Patients With Stage II or Stage III Cancer of the Larynx or Hypopharynx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aichi Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439499; AICHI-UHA-HN04-02
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Radiotherapy

INTERVENTIONS:
Drug: docetaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving docetaxel together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with radiation therapy works in treating patients with stage II or stage III cancer of the larynx or hypopharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response of the primary tumor in patients with stage II or III squamous cell carcinoma of the larynx or hypopharynx treated with docetaxel and radiotherapy.

Secondary

* Determine the local relapse-free survival of patients treated with this regimen.
* Determine the larynx-preservation survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the protocol completion rate in patients treated with this regimen.
* Determine the adverse effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on days 1, 8, 15, 22, and 29 and undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, and 29-33.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the larynx or hypopharynx

  * Stage II or III disease
* Solitary lymph node metastasis located in level II-III allowed
* Age 70 and over OR meets 1 of the following criteria:

  * Creatinine clearance 30-60 mL/min
  * History of platinum allergy
  * Diagnosis of unstable angina
  * Ineligible for systemic chemotherapy, including high-dose platinum-containing regimens

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Neutrophil count > 1,500/mm^3
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* AST and ALT ≤ 2.0 times upper limit of normal
* Bilirubin < 2.0 mg/dL
* No severe liver disease

Renal

* See Disease Characteristics
* Creatinine clearance ≥ 30 mL/min
* No severe renal disease

Pulmonary

* No severe pulmonary disease

Other

* No severe neurologic disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* No prior surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Objective response of primary tumor

SECONDARY OUTCOMES:
Local complete response rate
Local progression-free survival at 2 years
Local relapse-free survival
Larynx preservation survival at 2 years
Overall survival at 2 years
Treatment completion rate
Incidence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Nobukazu Fuwa, Study Chair — Aichi Cancer Center
Locations (9):
- Japan (9):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Hirosaki University, School of Medicine, Hirosaki, Aomori
  - Chiba University, Chiba, Chiba
  - Yokohama City University, Yokohama, Kanagawa
  - Shinshu University Health Center, Matsumoto, Nagano
  - Nara Medical University Cancer Center, Nara, Nara
  - Graduate School of Medical Science at the University of Ryukyu, Okinawa, Okinawa
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - National Hospital Organization - Medical Center of Kure, Hiroshima